CLINICAL TRIAL: NCT04167579
Title: The Society of Thoracic Surgeons and American College of Cardiology Foundation's Transcutaneous Valve Therapy (TVT) Registry
Brief Title: STS & ACC Foundation's Transcutaneous Valve Therapy (TVT) Registry Foundation's Transcutaneous Valve Therapy (TVT) Registry
Acronym: TVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Colleen Balius, CLINICAL DATA COORDINATOR (RN), Hoag Memorial Hospital Presbyterian
Other Study IDs: 172-19-CV
Record Dates: First submitted 2019-08-08; First posted 2019-11-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Transcutaneous Valve Therapies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcutaneous Valve Therapy — Any patient who undergoes an attempted transcutaneous aortic or mitral valve therapy procedure, with an FDA approved device.

SUMMARY:
The TVT Registry was designed to support a national surveillance system to assess the characteristics, treatments, and outcomes of patients receiving transcutaneous valve therapies.

DETAILED DESCRIPTION:
The TVT Registry was designed to support a national surveillance system to assess the characteristics, treatments, and outcomes of patients receiving transcutaneous valve therapies. Patient-level data are submitted by participating hospitals to The Society of Thoracic Surgeons (STS) and American College of Cardiology Foundation's (ACCF) joint TVT Registry. The purposes of the TVT Registry include: (i) collecting pertinent and standardized data elements from participating hospitals, health care providers and others that measure and assess the quality of care for patients receiving TVT; (ii) providing confidential periodic reports to participating hospitals, health care providers and others, to evaluate and improve the quality of care in these areas; and (iii) permitting and fostering appropriate research based upon the data collected by means of the TVT Registry.

The secondary aim of the TVT Registry is to serve as a scalable data infrastructure forpost market studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 and older) who undergo an attempted transcutaneous aortic or mitral valve therapy procedure, with an FDA approved device.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient who undergoes an attempted transcutaneous aortic or mitral valve therapy procedure, with an FDA approved device.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 30 days from procedure
  increase in the 30-day risk of adverse events among patients receiving TAVR

SECONDARY OUTCOMES:
Mortality | 1 year
  Proportion of patients who are alive with at least moderate functional improvement (defined as at least 10 point improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline) at 1 year after receiving TAVR
Major adverse cardiac and cerebrovascular events | 1 year from procedure
  increase in the 1 year risk of adverse events among patients receiving TAVR

CONTACTS AND LOCATIONS:
Locations (1):
- Hoah Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No